CLINICAL TRIAL: NCT07102602
Title: Feasibility of Assessing Muscle Displacement and Muscle Excursion on Muscle Fatigue, With and Without Preventive Strategies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 202410054DINE
Record Dates: First submitted 2025-07-31; First posted 2025-08-04 (Actual); Last update posted 2025-08-04 (Actual); Status verified 2025-07

CONDITIONS: Muscle Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- high intensity laser therapy (Active Comparator)
  Interventions: Device: high intensity laser therapy
- sham laser therapy (Sham Comparator)
  Interventions: Device: Sham laser therapy

INTERVENTIONS:
Device: high intensity laser therapy — The high-intensity laser used in this study is approved by the Ministry of Health and Welfare, Taiwan (No. 032670). It operates at a wavelength of 940 nm. For the active treatment (HILT), the laser delivers 900 joules to the quadriceps at a power output of 3 W for 5 minutes and is applied along the length of the quadriceps muscle
  Arms: high intensity laser therapy
Device: Sham laser therapy — In the sham condition (SHAM), the output is set to 0 W for 5 minutes, resulting in no energy delivery.
  Arms: sham laser therapy

SUMMARY:
Study Subjects: This study will recruit healthy males aged 18 to 35 who regularly exercise for at least 2.5 hours per week.

Expected Number of Participants: 20.

Methods and Procedures: This trial will be randomized into two groups, Groups A and B, who will undergo two isokinetic concentric exercise sessions (fatiguing exercise) separated by 15 days. Group A will first receive a fatigue prevention strategy (high-energy laser) followed by a placebo-controlled no-fatigue strategy 15 days later. Group B will first receive a placebo-controlled no-fatigue strategy followed by a fatigue prevention strategy (high-energy laser) 15 days later. The fatigue prevention strategy involves irradiating the quadriceps femoris with a 900-joule high-intensity laser therapy (3-watt output power for 5 minutes) before the isokinetic concentric exercise. The no-fatigue strategy (sham-controlled) involves irradiating the quadriceps femoris with a 0-joule high-energy laser (0-watt output power for 5 minutes) before the isokinetic concentric exercise. Muscle displacement, muscle excursion, as well as muscle electrophysiological changes, force output, and microcirculation parameters were measured before and after exercise to verify the feasibility of muscle displacement and migration for muscle fatigue assessment, and to further establish their impact and application value in muscle fatigue prevention strategies (high-intensity laser therapy).

ELIGIBILITY:
Inclusion Criteria:

* healthy male aged between 18 and 35 years who engage in regular physical activity for at least 2.5 hours per week

Exclusion Criteria:

* history of musculoskeletal injuries or lower limb muscle strains involving the dominant lower limb within the past six months
* history of surgical interventions on the dominant lower limb

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Muscle displacement | pre-fatigue (baseline), immediately post-fatigue, 5, 10, 20 minutes post-fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University College of Medicine, Taipei, Taipei city, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided